CLINICAL TRIAL: NCT04521569
Title: A Randomized, Blinded, Multi-site, Pilot Study to Evaluate Adenosine 2A Receptor Agonist (REGADENOSON) in the Rehabilitation of Marginal Donor Lungs.
Brief Title: Regadenoson Infusion of Marginalized Donor Lungs in an EVLP System
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Christine Lau, Surgeon-in-Chief, Department of Surgery, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UVA-LAU-02; 5R01HL128492-04 (NIH)
Record Dates: First submitted 2020-07-14; First posted 2020-08-20 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Lung Transplant
Keywords: EVLP; Lung Transplantation
MeSH Terms: interventions — regadenoson

STUDY DESIGN:
Intervention Model Description: Randomization to the EVLP with placebo or EVLP with Regadenoson groups will be performed in a 1:2 ratio.
Who Masked: Participant, Care Provider, Investigator
Masking Description: All study team members and subjects will be blinded to treatment assignment with the exception of the statisticians and investigational pharmacist preparing the study treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EVLP with Regadenoson (Experimental): Following the routine retrieval procedure of the lungs, they will be placed on the EVLP circuit (XVIVO Perfusion System) and infused with the study drug, Regadenoson.
  Interventions: Drug: Regadenoson
- EVLP with Steen solution (Placebo Comparator): Following the routine retrieval procedure of the lungs, they will be placed on the EVLP circuit (XVIVO Perfusion System) and infused with the same volume of Steen solution.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Regadenoson — If the donor lungs are randomized the experimental arm, the administration of Regadenoson will be performed at each study site by a qualified medical professional. The donor lungs will be perfused with Regadenoson at a dosage of 1.44 microgram/kg/min (based on donor's weight) for a minimum of three hours and maximum of four hours, using a pediatric syringe pump into the EVLP circuit (XVIVO Perfusion System). The infusion will begin within 10 minutes of the start of the EVLP procedure. Once the EVLP is complete the lungs are re-flushed with Perfadex solution (removing the Steen™ solution and Regadenoson; standard for EVLP).
  Other Names: Lexiscan
  Arms: EVLP with Regadenoson
Drug: Placebo — If the donor lungs are randomized to the Steen solution arm, the donor lungs will be perfused with placebo at a rate equivalent to the dosage of Regadenoson (1.44 microgram/kg/min), for a minimum of three hours and maximum of four hours, using the same pediatric syringe pump. The infusion will begin within 10 minutes of the start of the EVLP procedure.
  Other Names: Steen solution
  Arms: EVLP with Steen solution

SUMMARY:
The purpose of this study is to see if adding a drug called Regadenoson to the EVLP circulation reservoir during perfusion of marginal donor lungs will help increase the likelihood that the donor lungs will become usable for transplantation.

DETAILED DESCRIPTION:
Lung transplantation currently is one way to treat a variety of serious diseases and conditions such as emphysema, pulmonary fibrosis, and cystic fibrosis. Ischemia Reperfusion Injury (IRI) is a known problem that can happen during the first few days after a lung transplant. IRI can cause swelling of the lungs and low levels of oxygen. The most serious type of IRI can cause the transplanted lung to not work properly, it can even cause death. While new treatments and practices have been put into place to lower the chances of IRI, it is still a difficult problem to overcome after a lung transplant.

Molecule called Adenosine 2A receptor (A2AR) have been studied in animals with IRI for many years. Some of these studies suggest that with the use of A2AR agonist, the chance of IRI may be lowered or prevented. Regadenoson is a selective A2AR agonist.

ELIGIBILITY:
Inclusion Criteria:

Donor Lung Inclusion Criteria for EVLP

1. At the time of clinical evaluation, the PaO2/FiO2 ≤ 300mm Hg OR
2. If the PaO2/FiO2 is > 300mm hg and the donor has any one of more of the following donor risk factors:

   1. Multiple blood transfusions
   2. Pulmonary Edema detected via CXR, Bronchoscopy or palpation of the lungs
   3. Donation after cardiac death donors
   4. High risk donor history (example: asphyxia, hanging, drowning)

Donor lung Inclusion Criteria for Transplant Suitability after EVLP

1. Delta PaO2 greater than 350 mmhg (measured with an FiO2 set at 1.0) at two consecutive time periods at 2, 3, or 4 hours of EVLP.
2. Stability or improvement of other lung function parameters during EVLP perfusion, such as PVR, compliance, or airway pressures.
3. Lungs clinically suitable for transplantation (e.g. without signs of significant contusions, edema, or secretion) in the opinion of the surgical investigator(s).

Participant Inclusion Criteria

1. Subjects must be undergoing a single or bilateral lung transplantation for end-stage lung disease and thus meet all criteria to be listed. Single lungs are only allowable when initially placed as bilaterally block on EVLP circuit.
2. Male or female subject, 18 -75 years of age.
3. Subject agrees to accept EVLP perfused lungs.
4. Subjects must sign a study specific informed consent prior to study entry.

Exclusion Criteria:

Donor Lung Exclusion Criteria for EVLP

1. Donor lung has significant pneumonia as defined by positive bacterial growth in blood culture (not related to other source of infection) or persistent purulent, un-clearable secretions on bronchoscopy OR as determined by the investigator.
2. Donor has aspirated gastric contents into the lung. Donor lung has significant mechanical lung injury or trauma.
3. Donor lung has active infections disease, such as HIV, Hepatitis B or C, HTLV or syphilis.
4. Donor lung must not be split and perfused as single lung on EVLP circuit.

Donor Lung Exclusion Criteria for Transplant Suitability after EVLP (All of the below must be negative)

1. Delta PaO2 less than 350 mmHg (measured with FiO2 set at 1.0) at two consecutive time periods at 2, 3 or 4 hours of ex Vivo perfusion.
2. > 10% functional deterioration of other lung parameters during EVLP such as PVR, compliance or airway pressures.

Participant Exclusion Criteria

1. Subject requires preoperative extracorporeal membrane oxygenation (ECMO).
2. Subjects who are receiving or have received within 30 days any other investigational agents.
3. Subjects with Burkolderia cepacia.
4. Subjects who have had a previous lung transplant.
5. Subjects who have an uncontrolled concurrent illness including, but not limited to an ongoing or active infection, uncontrolled congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements per investigator discretion.
6. Pregnant or breastfeeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2024-06-23 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Lung Rehabilitation | 30 days
  The primary endpoint is rehabilitation (yes, no) for marginal donor lungs that undergo ex-vivo perfusion using a "lung box" as assessed by the transplant surgeon and utilizing the "Toronto Method" clinical protocol. Rate of rehabilitation is defined as the proportion of sets of lungs that underwent EVLP with/without Regadenoson treatment and are determined to be eligible for implant.

SECONDARY OUTCOMES:
Primary Lung Graft Dysfunction (PGD) Score | 72 hours
  Primary graft dysfunction (PGD) is a clinical entity that reflects the development of early acute lung injury after lung transplantation. PGD severity is graded between 0 and 3 and it is measured at 6h, 12h, 24h, 48h and 72 hours after lung transplantation. A score of Score 0 means no PGD and 1-3 increasingly more severe. 3 is so severe requires ECMO support.
Intensive care unit length of stay | 8 weeks
  Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
Using of ECMO | 1 week
  How often the patient will use ECMO due to lung infection after lung transplantation
Duration on ventilator post-Operative | 1 month
  Will measure how long the patient use ventilator post-operation.
12-month survival | 12 months
  Patient survival 360 days after lung transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Christine Lau, MD, Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - University of Maryland Medical Center, Baltimore, Maryland
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No